CLINICAL TRIAL: NCT07272564
Title: Periodontal Inflammation and Tryptophan-Kynurenine Metabolism in Parkinson's Disease
Brief Title: Kynurenine Pathway in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melis Yilmaz, Assistant Prof Dr, Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1082
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases; Inflammation
Keywords: periodontal disease; Tryptophan; Kynurenine
MeSH Terms: conditions — Periodontal Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Saliva and serum samples were collected from periodontitis patients and with Parkinson's +periodontitis patients. Samples were analyzed for TRP, KYN, KYN/TRP ratio, KYNA, 3OHKYN, picolinic acid (PA), and quinolinic acid (QA) by liquid chromatography-mass spectrometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Saliva and serum collection of patients and samples molecules analysis
  Interventions: Other: Saliva and serum sampling
- Experimental (Experimental): Samples were analyzed for TRP, KYN, KYN/TRP ratio, KYNA, 3OHKYN, picolinic acid (PA), and quinolinic acid (QA) by liquid chromatography-mass spectrometry. Clinical periodontal parameters [plaque index (PI), probing pocket depth (PPD), clinical attachment loss (CAL), and bleeding on probing (BOP)] were recorded.
  Interventions: Other: Saliva, serum and GCF sampling

INTERVENTIONS:
Other: Saliva and serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Arms: Active Comparator
Other: Saliva, serum and GCF sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Arms: Experimental

SUMMARY:
Parkinson's disease is a slowly progressing disease that affects the motor and non-motor functions of an individual. Periodontitis is an inflammatory chronic disease resulting in the destruction of tooth supporting structures. Inflammation has been identified as an important factor in both diseases. Given this common mechanism, the question arises as to how they may affect each other when both diseases occur together. In this study, we compared the metabolism of tryptophan, a natural amino acid of the human body, and observed whether such a process provides a biological link between periodontitis and Parkinson's disease. We extracted the saliva and blood samples of patients of Parkinson's disease and periodontitis, patients of periodontitis and healthy human beings. Comparisons between the three were made, and it was found that levels of some metabolites of tryptophan were higher in the patients of both diseases. These findings raise the possibility of a close biological connection between periodontal and brain health. Through an increased understanding of this connection in the future, new approaches for diagnosis and treatment of Parkinson's disease and periodontitis may be developed.

DETAILED DESCRIPTION:
Saliva and serum samples were collected from 20 Stage III, Grade B periodontitis patients with PAD (Parkinson+periodontitis group) and without PAD (periodontitis group), and 20 periodontally and systemically healthy (control group). Samples were analyzed for TRP, KYN, KYN/TRP ratio, KYNA, 3OHKYN, picolinic acid (PA), and quinolinic acid (QA) by liquid chromatography-mass spectrometry. Clinical periodontal parameters [plaque index (PI), probing pocket depth (PPD), clinical attachment loss (CAL), and bleeding on probing (BOP)] were recorded.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy

  * clinical diagnosis of periodontitis
  * clinical diagnosis of periodontal health

Exclusion Criteria:

* history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)

  * nonsurgical periodontal treatment (previous 6 months)
  * surgical periodontal treatment (previous 12 months)
  * presence of<10 teeth
  * current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
  * diabetes
  * diagnosis of rheumatoid arthritis
  * pregnancy
  * lactating
  * smoking
  * excessive alcohol consumption.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 6 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Saliva and serum samples processing and analyses | 1 month
  Samples were analyzed for TRP, KYN, KYN/TRP ratio, KYNA, 3OHKYN, picolinic acid (PA), and quinolinic acid (QA) by liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No